CLINICAL TRIAL: NCT02667210
Title: Retrospective Cohort Study to Evaluate the Relation Between Doctor/Pharmacy Shopping and Outcomes Suggestive of Misuse, Diversion, Abuse and/or Addiction by Medical Record Review
Brief Title: Study to Eval Relation Btw Doctor/Pharmacy Shopping & Outcomes of Misuse, Diversion, Abuse, Addiction by Med Rec Review
Status: Completed | Type: Observational
Sponsor: Member Companies of the Opioid PMR Consortium (Industry)
Collaborators: HealthCore, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Observational Study 3033-10; Study 3033-10 (Other: Member Companies of the Opioid PMR Consortium)
Record Dates: First submitted 2016-01-21; First posted 2016-01-28 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Opioid-Related Disorders; Opiate Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- No shopping behavior
  Interventions: Other: Medical Record Review
- Minimal shopping behavior
  Interventions: Other: Medical Record Review
- Marked shopping behavior
  Interventions: Other: Medical Record Review
- Extensive shopping behavior
  Interventions: Other: Medical Record Review

INTERVENTIONS:
Other: Medical Record Review — Medical Record Review of Behaviors Suggestive of Misuse, Diversion, Abuse and/or Addiction

SUMMARY:
To assess whether the percentage of patients with behaviors suggestive of misuse, diversion, abuse and/or addiction described in the medical record increases across pre-defined categories of increasing doctor/pharmacy shopping behavior.

DETAILED DESCRIPTION:
Based on a review of the literature, the Food and Drug Administration (FDA) concluded that more data are needed regarding the serious risks of misuse, abuse, addiction, overdose, and death associated with the long-term use of extended release/long acting (ER/LA) opioid analgesics. Thus, the FDA is requiring that ER/LA opioid analgesic drug sponsors conduct post-marketing studies to assess these risks. The four observational post-marketing requirement (PMR) studies are labeled Study #2065-1, Study #2065-2, Study #2065-3, and Study #2065-4.

The objective of PMR Study #2065-4 is to define and validate doctor/pharmacy shopping as outcomes suggestive of misuse, diversion, abuse and/or addiction.

Study #2065-4 consists of three sub-studies, Study 4A, Study 4B, and Study 4C. In the current study (#2065-4 sub-study, Study 4C), the association of doctor/pharmacy shopping behavior with misuse, diversion, abuse and/or addiction will be assessed by reviewing medical charts in a sample of patients within specific categories of a priori defined doctor/pharmacy shopping. The four categories of doctor/pharmacy shopping behaviors identified and defined in Study 4A and will be applied to Study 4C. The medical chart is a rich source of information about the patient's medical conditions and behaviors suggestive of misuse and abuse. Medical record review for behaviors suggestive of misuse and abuse in patients with chronic pain discriminates between patients with and without opioid use disorders. Therefore, Study 4C was designed to utilize an insurance/health plan database (HealthCore Integrated Research Database [HIRD]) with access to medical records, to evaluate the association of a priori defined categories of doctor/pharmacy shopping and behaviors suggestive of misuse, diversion, abuse and/or addiction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older on the date of first IR or ER/LA opioid dispensing in 2012
2. Patients with at least two dispensings of any IR or ER/LA opioid. The first of these dispensings will have occurred in 2012 and an additional dispensing within 18 months after the first.
3. Continuous, fully insured enrollment with medical and pharmacy eligibility in a health plan included in the HealthCore Integrated Research Database (HIRD) for at least six months prior to the start of the follow-up period.
4. Patients with continuous enrollment during the follow-up period of 18 months

Exclusion Criteria:

1. Patients who cannot be classified into one of the four a priori defined doctor/pharmacy shopping categories
2. Patients for whom no medical records can be accessed
3. Patients with a known history of abuse identified through the administrative claims data will be excluded because HealthCore is not permitted to request their medical records.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients identified from the HealthCore Integrated Research Database
Sampling Method: Probability Sample
Enrollment: 590 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
The percentages of patients in each category having at least one and up to 34 (all) of the prespecified list of behaviors suggestive of misuse, diversion, abuse and/or addiction in their medical records | Retrospective review over 24 month period starting 6 months prior to first dispensing in 2012 and 18 month follow-up
The correlation among the behaviors suggestive of misuse, diversion, abuse and/or addiction | Retrospective review over 24 month period starting 6 months prior to first dispensing in 2012 and 18 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Cepeda, MD, PhD, Study Chair — Janssen Research & Development, LLC